CLINICAL TRIAL: NCT03704792
Title: Validation of the Second Generation of the Controlled Attenuation Parameter (CAP) Using the MRI-PDFF as Reference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M134
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult CLD Group (Experimental): Only one group of patients in the study: adult patients with chronic liver disease (CLD), all etiologies combined, who will have a FibroScan 530 Compact examination to calculate the CAP value.
  Interventions: Device: FibroScan 530 Compact

INTERVENTIONS:
Device: FibroScan 530 Compact — The FibroScan® is a device equipped with probes (M+ or XL+), each of which consists of an ultrasonic transducer mounted on the axis of a mechanical vibrator. Liver stiffness and CAP measurements are performed on the right lobe of the liver with the patient in a dorsal decubitus and maximal abduction position. The procedure is non-invasive and painless.

SUMMARY:
Chronic liver diseases (CLDs) represent a major worldwide public health burden. Worldwide estimations show that 844 million people have CLDs, a lot more than other chronic diseases such as diabetes or cardiovascular diseases. CLD is most of the time an asymptomatic, progressive, and potentially fatal disease. With its complications it becomes one of the major causes of mortality worldwide. Globally, hepatitis B virus and hepatitis C virus, alcoholic liver disease and non-alcoholic steatohepatitis, are the most important causes of liver disease.

The diagnosis of liver lesions remains an important issue for these patients. The prognosis and management of liver disease greatly depends on the amount of liver fibrosis. In early stages, it is the main factor predicting long-term outcome of these patients. The liver biopsy still represents the gold standard diagnostic tool for liver fibrosis assessment, although a wide spectrum of noninvasive tools are now commonly used as a surrogate to the liver biopsy. It includes direct and indirect serum markers of liver fibrosis, but also several imaging-based methods, including transient elastography (FibroScan®, Echosens, Paris, France).

Even if the liver fibrosis is the key pathological feature of progressive liver disease, the accumulation of excessive hepatic triglyceride, hepatic steatosis, is today recognized as an important factor in the pathogenesis of a number of CLD. The magnetic resonance imaging (MRI) techniques are sensitive to steatosis and show interesting diagnostic performances, especially the MRI using the proton density fat fraction (MRI-PDFF) which has shown at least equivalence in accuracy for quantifying hepatic steatosis with both 1H Magnetic Resonance Spectroscopy and with histological grade, across several studies. Therefore, this technique is now part of the gold standard diagnostic tool to establish the grade of hepatic steatosis. Echosens has developed an ultrasonic controlled attenuation parameter (CAP) designed to quantify hepatic steatosis using a process based on vibration controlled transient elastography (VCTE™).

Echosens is working on improving the diagnostic accuracy of the CAP measurement performed with the FibroScan. This protocol is set-up to compare the diagnostic performances of the first generation of the CAP and the second generation of the CAP to the reference, the MRI-PDFF, in patients with CLD, all etiologies combined.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years of age
* Patient must be able to give written informed consent
* Patient affiliated to a social security system
* Patient with a chronic liver disease, all etiologies

Exclusion Criteria:

* Vulnerable patient
* Pregnant women
* Patient with presence of ascites
* Contra-indication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Liver fat content assessed by MRI-PDFF. | 12 months

SECONDARY OUTCOMES:
Ratio IQR CAPv1/CAPv2 and/or ratio standard deviation CAPv1/CAPv2 | 12 months
Difference between CAPv1 and CAPv2 measures | 12 months
Correlation between CAPv1, CAPv2 and MRI-PDFF | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpitaux Universitaires Paris Seine Saint-Denis - Service Hépatologie, Bondy
  - Centre Hospitalier Universitaire de Bordeaux - Hôpital Haut Lévêque, Bordeaux
  - Hôpital Saint-Antoine - Service Hépatologie, Paris
  - CHU Rennes Hôpital Pontchaillou - Service des Maladies du Foie, Rennes

IPD SHARING:
Plan to Share IPD: Undecided